CLINICAL TRIAL: NCT01682083
Title: COMBI-AD: A Phase III Randomized Double Blind Study of Dabrafenib (GSK2118436) in COMBInation With Trametinib (GSK1120212) Versus Two Placebos in the ADjuvant Treatment of High-risk BRAF V600 Mutation-positive Melanoma After Surgical Resection
Brief Title: Dabrafenib With Trametinib in the Adjuvant Treatment of High-risk BRAF V600 Mutation-positive Melanoma (COMBI-AD).
Acronym: COMBI-AD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 115532; 2012-001266-15 (EudraCT Number); CDRB436F2301 (Other: Novartis)
Record Dates: First submitted 2012-09-06; First posted 2012-09-10 (Estimated); Results first posted 2018-09-26 (Actual); Last update posted 2023-08-30 (Actual); Status verified 2023-08

CONDITIONS: Melanoma
Keywords: MEK inhibitor; trametinib; Oncology; adjuvant melanoma; dabrafenib; dabrafenib and trametinib combination therapy; BRAF mutation-positive melanoma; BRAF inhibitor
MeSH Terms: conditions — Melanoma; Neoplasms | interventions — dabrafenib; trametinib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dabrafenib and trametinib (Experimental): Subjects received dabrafenib (150 mg twice daily) and trametinib (2 mg once daily) orally for 12 months.
  Interventions: Drug: Dabrafenib; Drug: Trametinib
- Dabrafenib and trametinib placebos (Placebo Comparator): Subjects received matching placebos orally for 12 months
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Dabrafenib — Each capsule contained 50 mg or 75 mg of free base (present as the mesylate salt)
  Other Names: GSK2118436
  Arms: Dabrafenib and trametinib
Drug: Trametinib — Each tablet contained 0.5 mg or 2.0 mg of trametinib parent (present as the DMSO solvate)
  Other Names: GSK1120212
  Arms: Dabrafenib and trametinib
Drug: Placebos — The placebo capsules and tablets contained the same inactive ingredients and film coatings as the dabrafenib and trametinib study treatment
  Arms: Dabrafenib and trametinib placebos

SUMMARY:
This was a two-arm, randomized, double-blind Phase III study of dabrafenib in combination with trametinib versus two placebos in the adjuvant treatment of melanoma after surgical resection. Patients with completely resected, histologically confirmed, BRAF V600E/K mutation-positive, high-risk [Stage IIIa (lymph node metastasis >1 mm), IIIb or IIIc] cutaneous melanoma were screened for eligibility. Subjects were randomized to receive either dabrafenib (150 milligram (mg) twice daily [BID]) and trametinib (2 mg once daily [QD]) combination therapy or two placebos for 12 months.

DETAILED DESCRIPTION:
This was a two-arm, randomized, double-blind, multi-center, international phase III study of dabrafenib in combination with trametinib versus two matching placebos in the adjuvant treatment of melanoma after surgical resection. Patients with completely resected, histologically confirmed, BRAF V600E/K mutation-positive, high-risk [Stage IIIa (lymph node metastasis >1 mm), IIIb or IIIc] cutaneous melanoma were screened for eligibility. Subjects were randomized to receive either dabrafenib (150 milligram (mg) twice daily [BID]) and trametinib (2 mg once daily [QD]). None of the patients had undergone previous systemic anticancer treatment or radiotherapy for melanoma. All the patients had undergone completion lymphadenectomy with no clinical or radiographic evidence of residual regional node disease within 12 weeks before randomization, had recovered from definitive surgery, and had an Eastern Cooperative Oncology Group performance status of 0 or 1. BRAF V600 mutation status was confirmed in primary-tumor or lymph-node tissue by a central reference laboratory. All the patients provided written informed consent.

The primary end point was recurrence-free survival, Overall survival, as the key secondary end point, was to be tested in a hierarchical manner only if the primary end point met the criteria for significance. The overall survival analysis used a preplanned three-look Lan-DeMets group sequential design with an O'Brien-Fleming-type boundary, which was used to determine the significance threshold for the first interim overall survival analysis (two-sided P=0.000019).

Disease assessments included clinical examination and imaging by means of computed tomography, magnetic resonance imaging, or both.) Imaging was performed every 3 months during the first 24 months, then every 6 months until disease recurrence or the completion of the trial. Follow-up for survival began after recurrence and continued through the end of the trial. Adverse events and laboratory values were assessed at screening, on the date of randomization, at least once per month through month 12, and at every visit for disease-recurrence assessment after month 12. Adverse events and laboratory values were graded according to the Common Terminology Criteria for Adverse Events, version 4.0.

ELIGIBILITY:
Key Inclusion Criteria:

* Completely resected histologically confirmed high-risk [Stage IIIa (LN metastasis more than 1 mm), IIIb or IIIc cutaneous melanoma determined to be V600E/K mutation positive by a central laboratory. Patients presenting with initial resectable lymph node recurrence after a diagnosis of Stage I or II melanoma are eligible.
* Surgically rendered free of disease no more than 12 weeks before randomization.
* Recovered from definitive surgery (e.g. no uncontrolled wound infections or indwelling drains).
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-1.
* Adequate hematologic, hepatic, renal and cardiac function.

Key Exclusion Criteria:

* Known mucosal or ocular melanoma or the presence of unresectable in-transit metastases.
* Evidence of distant metastatic disease.
* Prior systemic anti-cancer treatment and radiotherapy for melanoma; prior surgery for melanoma is allowed.
* History of another malignancy or concurrent malignancy including prior malignant melanoma. Exceptions to this include: Patients who have been disease-free for 5 years or patients with a history completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible, for example cervical cancer in situ, atypical melanocytic hyperplasia or melanoma in situ, multiple primary melanomas, or other malignancies for which the patient has been disease free for > 5 years.
* History or current evidence of cardiovascular risk.
* History or current evidence of retinal vein occlusion (RVO) or central serous retinopathy (CSR)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 870 (Actual)
Dates: Start 2013-01-08 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2023-07-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (187):
- United States (27):
  - Novartis Investigative Site, Birmingham, Alabama
  - Novartis Investigative Site, Tucson, Arizona
  - Novartis Investigative Site, San Francisco, California
  - Novartis Investigative Site, Aurora, Colorado
  - Novartis Investigative Site, Farmington, Connecticut
  - Novartis Investigative Site, Fort Myers, Florida
  - Novartis Investigative Site, Lake Worth, Florida
  - Novartis Investigative Site, Orlando, Florida
  - Novartis Investigative Site, St. Petersburg, Florida
  - Novartis Investigative Site, Stuart, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Baltimore, Maryland
  - Novartis Investigative Site, Lutherville-Timonium, Maryland
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Ann Arbor, Michigan
  - Novartis Investigative Site, Morristown, New Jersey
  - Novartis Investigative Site, Winston-Salem, North Carolina
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Dallas, Texas
  - Novartis Investigative Site, Murray, Utah
  - Novartis Investigative Site, Seattle, Washington
- Argentina (6):
  - Novartis Investigative Site, Capital Federal, Buenos Aires
  - Novartis Investigative Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Novartis Investigative Site, Viedma, Río Negro Province
  - Novartis Investigative Site, Rosario, Santa Fe Province
  - Novartis Investigative Site, Buenos Aires
  - Novartis Investigative Site, Santa Fe
- Australia (12):
  - Novartis Investigative Site, Gateshead, New South Wales
  - Novartis Investigative Site, North Sydney, New South Wales
  - Novartis Investigative Site, Tweed Heads, New South Wales
  - Novartis Investigative Site, Westmead, New South Wales
  - Novartis Investigative Site, Greenslopes, Queensland
  - Novartis Investigative Site, Milton, Queensland
  - Novartis Investigative Site, Woolloongabba, Queensland
  - Novartis Investigative Site, Adelaide, South Australia
  - Novartis Investigative Site, Box Hill, Victoria
  - Novartis Investigative Site, Heidelberg, Victoria
  - Novartis Investigative Site, Melbourne, Victoria
  - Novartis Investigative Site, Nedlands, Western Australia
- Austria (6):
  - Novartis Investigative Site, Graz
  - Novartis Investigative Site, Innsbruck
  - Novartis Investigative Site, Linz
  - Novartis Investigative Site, Salzburg
  - Novartis Investigative Site, Vienna
  - Novartis Investigative Site, Wels
- Belgium (4):
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Leuven
  - Novartis Investigative Site, Liège
  - Novartis Investigative Site, Wilrijk
- Brazil (5):
  - Novartis Investigative Site, Goiânia, Goiás
  - Novartis Investigative Site, Curitiba, Paraná
  - Novartis Investigative Site, Ijuí, Rio Grande do Sul
  - Novartis Investigative Site, Rio de Janeiro
  - Novartis Investigative Site, São Paulo
- Canada (7):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Hamilton, Ontario
  - Novartis Investigative Site, Oshawa, Ontario
  - Novartis Investigative Site, Ottawa, Ontario
  - Novartis Investigative Site, Toronto, Ontario
  - Novartis Investigative Site, Montreal, Quebec
  - Novartis Investigative Site, Québec, Quebec
- Czechia (5):
  - Novartis Investigative Site, Brno
  - Novartis Investigative Site, Hradec Králové
  - Novartis Investigative Site, Olomouc
  - Novartis Investigative Site, Prague
  - Novartis Investigative Site, Zlín
- Denmark (3):
  - Novartis Investigative Site, Arhus C
  - Novartis Investigative Site, Herlev
  - Novartis Investigative Site, Odense
- France (16):
  - Novartis Investigative Site, Bordeaux
  - Novartis Investigative Site, Boulogne-Billancourt
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, Dijon
  - Novartis Investigative Site, Grenoble
  - Novartis Investigative Site, Lille
  - Novartis Investigative Site, Marseille
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Nice
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Pierre-Bénite
  - Novartis Investigative Site, Reims
  - Novartis Investigative Site, Rennes
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Tours
  - Novartis Investigative Site, Villejuif
- Germany (32):
  - Novartis Investigative Site, Freiburg im Breisgau, Baden-Wurttemberg
  - Novartis Investigative Site, Heidelberg, Baden-Wurttemberg
  - Novartis Investigative Site, Heilbronn, Baden-Wurttemberg
  - Novartis Investigative Site, Mannheim, Baden-Wurttemberg
  - Novartis Investigative Site, Tübingen, Baden-Wurttemberg
  - Novartis Investigative Site, Ulm, Baden-Wurttemberg
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Nuremberg, Bavaria
  - Novartis Investigative Site, Regensburg, Bavaria
  - Novartis Investigative Site, Würzburg, Bavaria
  - Novartis Investigative Site, Darmstadt, Hesse
  - Novartis Investigative Site, Kassel, Hesse
  - Novartis Investigative Site, Marburg, Hesse
  - Novartis Investigative Site, Wiesbaden, Hesse
  - Novartis Investigative Site, Buxtehude, Lower Saxony
  - Novartis Investigative Site, Hanover, Lower Saxony
  - Novartis Investigative Site, Schwerin, Mecklenburg-Vorpommern
  - Novartis Investigative Site, Aachen, North Rhine-Westphalia
  - Novartis Investigative Site, Bochum, North Rhine-Westphalia
  - Novartis Investigative Site, Bonn, North Rhine-Westphalia
  - Novartis Investigative Site, Cologne, North Rhine-Westphalia
  - Novartis Investigative Site, Essen, North Rhine-Westphalia
  - Novartis Investigative Site, Münster, North Rhine-Westphalia
  - Novartis Investigative Site, Mainz, Rhineland-Palatinate
  - Novartis Investigative Site, Homburg, Saarland
  - Novartis Investigative Site, Magdeburg, Saxony-Anhalt
  - Novartis Investigative Site, Quedlinburg, Saxony-Anhalt
  - Novartis Investigative Site, Kiel, Schleswig-Holstein
  - Novartis Investigative Site, Lübeck, Schleswig-Holstein
  - Novartis Investigative Site, Erfurt, Thuringia
  - Novartis Investigative Site, Gera, Thuringia
  - Novartis Investigative Site, Berlin
- Greece (2):
  - Novartis Investigative Site, Athens
  - Novartis Investigative Site, Thessaloniki
- Israel (2):
  - Novartis Investigative Site, Jerusalem
  - Novartis Investigative Site, Ramat Gan
- Italy (7):
  - Novartis Investigative Site, Rome, Lazio
  - Novartis Investigative Site, Genoa, Liguria
  - Novartis Investigative Site, Bergamo, Lombardy
  - Novartis Investigative Site, Milan, Lombardy
  - Novartis Investigative Site, Candiolo, Piedmont
  - Novartis Investigative Site, Pisa, Tuscany
  - Novartis Investigative Site, Padua, Veneto
- Japan (2):
  - Novartis Investigative Site, Shizuoka
  - Novartis Investigative Site, Tokyo
- Netherlands (6):
  - Novartis Investigative Site, Amsterdam
  - Novartis Investigative Site, Groningen
  - Novartis Investigative Site, Leeuwarden
  - Novartis Investigative Site, Maastricht
  - Novartis Investigative Site, Nijmegen
  - Novartis Investigative Site, Rotterdam
- Novartis Investigative Site, Auckland, New Zealand
- Norway (2):
  - Novartis Investigative Site, Ålesund
  - Novartis Investigative Site, Oslo
- Poland (4):
  - Novartis Investigative Site, Gdansk
  - Novartis Investigative Site, Konin
  - Novartis Investigative Site, Poznan
  - Novartis Investigative Site, Warsaw
- Russia (5):
  - Novartis Investigative Site, Chelyabinsk
  - Novartis Investigative Site, Moscow
  - Novartis Investigative Site, Ryazan
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Volgograd
- Spain (12):
  - Novartis Investigative Site, Badalona
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Cartagena
  - Novartis Investigative Site, Donostia / San Sebastian
  - Novartis Investigative Site, Las Palmas de Gran Canaria
  - Novartis Investigative Site, Madrid
  - Novartis Investigative Site, Málaga
  - Novartis Investigative Site, Palma de Mallorca
  - Novartis Investigative Site, Pamplona
  - Novartis Investigative Site, Santander
  - Novartis Investigative Site, Seville
  - Novartis Investigative Site, Valencia
- Sweden (4):
  - Novartis Investigative Site, Gothenburg
  - Novartis Investigative Site, Lund
  - Novartis Investigative Site, Stockholm
  - Novartis Investigative Site, Uppsala
- Switzerland (3):
  - Novartis Investigative Site, Basel
  - Novartis Investigative Site, Chur
  - Novartis Investigative Site, Zurich
- Taiwan (3):
  - Novartis Investigative Site, Taichung
  - Novartis Investigative Site, Taipei
  - Novartis Investigative Site, Taoyuan District
- United Kingdom (11):
  - Novartis Investigative Site, Northwood, Middlesex
  - Novartis Investigative Site, Exeter
  - Novartis Investigative Site, Glasgow
  - Novartis Investigative Site, Guildford
  - Novartis Investigative Site, Leeds
  - Novartis Investigative Site, London
  - Novartis Investigative Site, Manchester
  - Novartis Investigative Site, Newcastle upon Tyne
  - Novartis Investigative Site, Norwich
  - Novartis Investigative Site, Preston
  - Novartis Investigative Site, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Syeda MM, Long GV, Garrett J, Atkinson V, Santinami M, Schadendorf D, Hauschild A, Millward M, Mandala M, Chiarion-Sileni V, Smylie M, Manikhas GM, Dummer R, Wiggins JM, Ali S, Adnaik SB, Tan M, Dajee M, Polsky D. Clinical validation of droplet digital PCR assays in detecting BRAFV600-mutant circulating tumour DNA as a prognostic biomarker in patients with resected stage III melanoma receiving adjuvant therapy (COMBI-AD): a biomarker analysis from a double-blind, randomised phase 3 trial. Lancet Oncol. 2025 May;26(5):641-653. doi: 10.1016/S1470-2045(25)00139-1. Epub 2025 Apr 15. PMID 40250457
- [Derived] Long GV, Hauschild A, Santinami M, Kirkwood JM, Atkinson V, Mandala M, Merelli B, Sileni VC, Nyakas M, Haydon A, Dutriaux C, Robert C, Mortier L, Schachter J, Schadendorf D, Lesimple T, Plummer R, Larkin J, Tan M, Adnaik SB, Burgess P, Jandoo T, Dummer R. Final Results for Adjuvant Dabrafenib plus Trametinib in Stage III Melanoma. N Engl J Med. 2024 Nov 7;391(18):1709-1720. doi: 10.1056/NEJMoa2404139. Epub 2024 Jun 19. PMID 38899716
- [Derived] Li SN, Wan X, Peng LB, Li YM, Li JH. Cost-effectiveness of immune checkpoint inhibition and targeted treatment in combination as adjuvant treatment of patient with BRAF-mutant advanced melanoma. BMC Health Serv Res. 2023 Jan 18;23(1):49. doi: 10.1186/s12913-023-09058-7. PMID 36653848
- [Derived] Schadendorf D, Robert C, Dummer R, Flaherty KT, Tawbi HA, Menzies AM, Banerjee H, Lau M, Long GV. Pyrexia in patients treated with dabrafenib plus trametinib across clinical trials in BRAF-mutant cancers. Eur J Cancer. 2021 Aug;153:234-241. doi: 10.1016/j.ejca.2021.05.005. Epub 2021 Jul 2. PMID 34225229
- [Derived] Dummer R, Hauschild A, Santinami M, Atkinson V, Mandala M, Kirkwood JM, Chiarion Sileni V, Larkin J, Nyakas M, Dutriaux C, Haydon A, Robert C, Mortier L, Schachter J, Lesimple T, Plummer R, Dasgupta K, Gasal E, Tan M, Long GV, Schadendorf D. Five-Year Analysis of Adjuvant Dabrafenib plus Trametinib in Stage III Melanoma. N Engl J Med. 2020 Sep 17;383(12):1139-1148. doi: 10.1056/NEJMoa2005493. Epub 2020 Sep 2. PMID 32877599
- [Derived] Dummer R, Brase JC, Garrett J, Campbell CD, Gasal E, Squires M, Gusenleitner D, Santinami M, Atkinson V, Mandala M, Chiarion-Sileni V, Flaherty K, Larkin J, Robert C, Kefford R, Kirkwood JM, Hauschild A, Schadendorf D, Long GV. Adjuvant dabrafenib plus trametinib versus placebo in patients with resected, BRAFV600-mutant, stage III melanoma (COMBI-AD): exploratory biomarker analyses from a randomised, phase 3 trial. Lancet Oncol. 2020 Mar;21(3):358-372. doi: 10.1016/S1470-2045(20)30062-0. Epub 2020 Jan 30. PMID 32007138
- [Derived] Schadendorf D, Hauschild A, Santinami M, Atkinson V, Mandala M, Chiarion-Sileni V, Larkin J, Nyakas M, Dutriaux C, Haydon A, Robert C, Mortier L, Lesimple T, Plummer R, Schachter J, Dasgupta K, Manson S, Koruth R, Mookerjee B, Kefford R, Dummer R, Kirkwood JM, Long GV. Patient-reported outcomes in patients with resected, high-risk melanoma with BRAFV600E or BRAFV600K mutations treated with adjuvant dabrafenib plus trametinib (COMBI-AD): a randomised, placebo-controlled, phase 3 trial. Lancet Oncol. 2019 May;20(5):701-710. doi: 10.1016/S1470-2045(18)30940-9. Epub 2019 Mar 27. PMID 30928620
- [Derived] Hauschild A, Dummer R, Schadendorf D, Santinami M, Atkinson V, Mandala M, Chiarion-Sileni V, Larkin J, Nyakas M, Dutriaux C, Haydon A, Robert C, Mortier L, Schachter J, Lesimple T, Plummer R, Dasgupta K, Haas T, Shilkrut M, Gasal E, Kefford R, Kirkwood JM, Long GV. Longer Follow-Up Confirms Relapse-Free Survival Benefit With Adjuvant Dabrafenib Plus Trametinib in Patients With Resected BRAF V600-Mutant Stage III Melanoma. J Clin Oncol. 2018 Dec 10;36(35):3441-3449. doi: 10.1200/JCO.18.01219. Epub 2018 Oct 22. PMID 30343620
- [Derived] Long GV, Hauschild A, Santinami M, Atkinson V, Mandala M, Chiarion-Sileni V, Larkin J, Nyakas M, Dutriaux C, Haydon A, Robert C, Mortier L, Schachter J, Schadendorf D, Lesimple T, Plummer R, Ji R, Zhang P, Mookerjee B, Legos J, Kefford R, Dummer R, Kirkwood JM. Adjuvant Dabrafenib plus Trametinib in Stage III BRAF-Mutated Melanoma. N Engl J Med. 2017 Nov 9;377(19):1813-1823. doi: 10.1056/NEJMoa1708539. Epub 2017 Sep 10. PMID 28891408

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 169 centers across 25 countries. Results reported have the data cut-off as of 30 June 2017.
Pre-assignment Details: Patients with completely resected, histologically confirmed, BRAF V600E/K mutation-positive, high-risk [Stage IIIA (lymph node metastasis >1 mm), IIIB, or IIIC] cutaneous melanoma.
Groups:
- Dabrafenib and Trametinib Combination Therapy: Subjects received dabrafenib (150 mg twice daily) and trametinib (2 mg once daily) orally for 12 months.
Period: Overall Study
Arm/Group | Dabrafenib and Trametinib Combination Therapy | Dabrafenib and Trametinib Placebos
Started | 438 | 432
Completed | 331 (Ongoing patients at the time of data cut-off. 3 patients were untreated) | 277 (Ongoing patients at the time of data cut-off.)
Not Completed | 107 | 155
Not completed — Lost to Follow-up | 11 | 18
Not completed — Withdrawal by Subject | 31 | 40
Not completed — Death | 60 | 93
Not completed — Physician Decision | 5 | 4

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat Population (ITT) consisted of all randomized patients whether or not randomized treatment was administered.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dabrafenib and Trametinib Combination Therapy | Dabrafenib and Trametinib Placebos | Total
Number analyzed (Participants) | 438 | 432 | 870
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.4 (14.17) | 50.5 (13.14) | 50.4 (13.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 195 | 193 | 388
  Male | 243 | 239 | 482
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 432 | 427 | 859
  Asian | 6 | 5 | 11

OUTCOME MEASURES:

1. Primary Outcome: Relapse-free Survival (RFS)
Description: Recurrence-free survival was defined as the time from randomization to disease recurrence (local recurrence, distant recurrence, second primary melanoma), or death from any cause.
Time Frame: Approximately 3.5 years
Population: Intent-to-Treat (ITT) Population
Measure: Number; unit: Participants with events
Arm/Group | Dabrafenib and Trametinib Combination Therapy | Dabrafenib and Trametinib Placebos
Number analyzed (Participants) | 438 | 432
Participants with events
  Relapsed (event) | 163 | 247
  Died | 3 | 1
  Censored, follow-up ended | 43 | 35
  Censored, follow-up ongoing | 229 | 149
Statistical Analysis 1: Comparison: Dabrafenib and Trametinib Combination Therapy vs Dabrafenib and Trametinib Placebos; The null hypothesis, H0: λ = 1 or reject it in favor of the alternative hypothesis, HA: λ ≠ 1, where λ is the hazard ratio (HR) of combination therapy relative to placebo; Test type: Superiority — Hazard ratio is obtained from the stratified Pike estimator. A hazard ratio <1 indicates a lower risk with Dabrafenib + Trametinib compared with Placebo; p < 0.0001, Log Rank; Hazard Ratio, log = 0.47, 95% CI 2-sided [0.39 to 0.58]

2. Secondary Outcome: Overall Survival
Description: Overall survival (OS) of dabrafenib and trametinib as a combination therapy versus placebo
Time Frame: approximately 3.5 years
Population: ITT population
Measure: Count of Participants; unit: Participants
Arm/Group | Dabrafenib and Trametinib Combination Therapy | Dabrafenib and Trametinib Placebos
Number analyzed (Participants) | 438 | 432
Participants
  Died (event) | 60 | 93
  Censored, follow-up ended | 47 | 62
  Censored, follow-up ongoing | 331 | 277
Statistical Analysis 1: Comparison: Dabrafenib and Trametinib Combination Therapy vs Dabrafenib and Trametinib Placebos; Hazard ratio is obtained from the stratified Pike estimator; Test type: Superiority — A hazard ratio <1 indicates a lower risk with dabrafenib + trametinib compared with Placebo; p = 0.006, Log Rank; the two-sided threshold for significance at this first interim analysis was p=0.000019; Hazard Ratio, log = 0.57, 95% CI 2-sided [0.42 to 0.79]

3. Secondary Outcome: Distant Metastasis-free Survival
Description: Distant metastasis-free survival (DMFS) of dabrafenib and trametinib as a combination therapy versus placebo. In the DMFS analysis, the first occurrence of distant metastasis or death (if it occurred before documented recurrence) was counted as an event.
Time Frame: approximately 3.5 years
Population: ITT population
Measure: Number; unit: Participants with events
Arm/Group | Dabrafenib and Trametinib Combination Therapy | Dabrafenib and Trametinib Placebos
Number analyzed (Participants) | 438 | 432
Participants with events
  Number of Subjects - Relapsed | 106 | 150
  Number of Subjects - died | 4 | 2
  Number of Subjects - censored, follow-up ended | 99 | 131
  Number of Subjects - follow-up ongoing | 229 | 149
Statistical Analysis 1: Comparison: Dabrafenib and Trametinib Combination Therapy vs Dabrafenib and Trametinib Placebos; Hazard ratio is estimated using Pike estimator; Test type: Superiority — A hazard ratio <1 indicates a lower risk with Dabrafenib + Trametinib compared with Placebo; Hazard Ratio, log = 0.51, 95% CI 2-sided [0.40 to 0.65]

4. Secondary Outcome: Freedom From Relapse
Description: Freedom from relapse (FFR) of dabrafenib and trametinib as a combination therapy versus placebo. In the FFR analysis, local or distant recurrence or a new primary melanoma were counted as events, and patients who died of causes other than melanoma or treatment-related toxicity were censored.
Time Frame: approximately 3.5 years
Population: ITT population
Measure: Number; unit: Participants with events
Arm/Group | Dabrafenib and Trametinib Combination Therapy | Dabrafenib and Trametinib Placebos
Number analyzed (Participants) | 438 | 432
Participants with events
  Number of Subjects - relapsed | 163 | 247
  Number of Subjects - died | 2 | 0
  Number of Subjects - censored, follow-up ended | 44 | 36
  Number of Subjects - censored, follow-up ongoing | 229 | 149
Statistical Analysis 1: Comparison: Dabrafenib and Trametinib Combination Therapy vs Dabrafenib and Trametinib Placebos; Hazard ratio is estimated using Pike estimator; Test type: Superiority — A hazard ratio <1 indicates a lower risk with Dabrafenib + Trametinib compared with Placebo; Hazard Ratio (HR) = 0.47, 95% CI 2-sided [0.39 to 0.57]

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from the time the first dose of study treatment is administered until 30 days after discontinuation of study treatment. Serious AEs (SAEs) were reported over the same time period as AEs except SAEs assessed as related to study participation, study treatment or concomitant medication were recorded from the time a subject consents to participate in the study up to and including any follow-up contact.
Description: All cause mortality provided for the treatment period only.
Groups:
- Dabrafenib + Trametinib Combination Therapy: Subjects received dabrafenib (150 mg twice daily) and trametinib (2 mg once daily) orally for 12 months.
Arm/Group | Dabrafenib + Trametinib Combination Therapy | Dabrafenib and Trametinib Placebos
All-Cause Mortality (participants affected / at risk) | 4/435 | 1/432
Serious Adverse Events (participants affected / at risk) | 155/435 | 44/432
Other Adverse Events (participants affected / at risk) | 414/435 | 340/432
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dabrafenib + Trametinib Combination Therapy (N=435) | Dabrafenib and Trametinib Placebos (N=432)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Pancytopenia (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Cardiac ventricular thrombosis (Cardiac disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 0 | 1
Chorioretinopathy (Eye disorders) | 5 | 0
Iritis (Eye disorders) | 1 | 0
Macular oedema (Eye disorders) | 1 | 0
Retinal detachment (Eye disorders) | 2 | 0
Uveitis (Eye disorders) | 2 | 0
Visual acuity reduced (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Pancreatic toxicity (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 0 | 1
Retroperitoneal haematoma (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 4 | 0
Asthenia (General disorders) | 1 | 0
Chills (General disorders) | 13 | 0
Fatigue (General disorders) | 2 | 0
Influenza like illness (General disorders) | 3 | 0
Pyrexia (General disorders) | 67 | 4
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0
Hepatic haemorrhage (Hepatobiliary disorders) | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 0
Abscess jaw (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 5 | 1
Cholecystitis infective (Infections and infestations) | 1 | 0
Epstein-Barr virus infection (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 8 | 1
Febrile infection (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Groin abscess (Infections and infestations) | 1 | 0
Groin infection (Infections and infestations) | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 1
Influenza (Infections and infestations) | 2 | 0
Lower respiratory tract infection (Infections and infestations) | 3 | 0
Parvovirus infection (Infections and infestations) | 1 | 0
Pharyngitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 3 | 0
Post procedural infection (Infections and infestations) | 0 | 1
Rash pustular (Infections and infestations) | 1 | 0
Retinitis (Infections and infestations) | 1 | 0
Salpingitis (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 4 | 0
Soft tissue infection (Infections and infestations) | 0 | 1
Subcutaneous abscess (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1
Urosepsis (Infections and infestations) | 1 | 0
Vulval abscess (Infections and infestations) | 1 | 0
Wound infection (Infections and infestations) | 0 | 1
Limb injury (Injury, poisoning and procedural complications) | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Seroma (Injury, poisoning and procedural complications) | 1 | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 3 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0
Blood creatine phosphokinase increased (Investigations) | 1 | 0
Ejection fraction decreased (Investigations) | 13 | 5
Right ventricular systolic pressure increased (Investigations) | 0 | 1
Transaminases increased (Investigations) | 1 | 0
Troponin increased (Investigations) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 0
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 2 | 0
Acanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Focal nodular hyperplasia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Keratoacanthoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Lentigo maligna (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 3
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Salivary gland adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 3
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1
Demyelinating polyneuropathy (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 2 | 0
Facial paralysis (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 4 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Meningoradiculitis (Nervous system disorders) | 1 | 0
Migraine (Nervous system disorders) | 1 | 1
Paraesthesia (Nervous system disorders) | 1 | 0
Peripheral sensorimotor neuropathy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 2 | 0
Seizure (Nervous system disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Obsessive-compulsive disorder (Psychiatric disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 0
Calculus urinary (Renal and urinary disorders) | 1 | 0
Nephrotic syndrome (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 1 | 0
Ovarian disorder (Reproductive system and breast disorders) | 1 | 0
Priapism (Reproductive system and breast disorders) | 1 | 0
Testicular mass (Reproductive system and breast disorders) | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 | 0
Panniculitis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash generalised (Skin and subcutaneous tissue disorders) | 1 | 0
Embolism (Vascular disorders) | 0 | 1
Hypotension (Vascular disorders) | 6 | 0
Lymphoedema (Vascular disorders) | 0 | 1
Vascular occlusion (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dabrafenib + Trametinib Combination Therapy (N=435) | Dabrafenib and Trametinib Placebos (N=432)
Neutropenia (Blood and lymphatic system disorders) | 34 | 4
Dry eye (Eye disorders) | 22 | 13
Vision blurred (Eye disorders) | 27 | 16
Abdominal pain (Gastrointestinal disorders) | 34 | 23
Abdominal pain upper (Gastrointestinal disorders) | 30 | 27
Constipation (Gastrointestinal disorders) | 51 | 27
Diarrhoea (Gastrointestinal disorders) | 143 | 65
Dry mouth (Gastrointestinal disorders) | 41 | 15
Dyspepsia (Gastrointestinal disorders) | 24 | 26
Nausea (Gastrointestinal disorders) | 172 | 88
Vomiting (Gastrointestinal disorders) | 120 | 43
Asthenia (General disorders) | 58 | 42
Chills (General disorders) | 158 | 19
Fatigue (General disorders) | 204 | 122
Influenza like illness (General disorders) | 66 | 29
Oedema peripheral (General disorders) | 58 | 19
Pyrexia (General disorders) | 248 | 44
Folliculitis (Infections and infestations) | 24 | 9
Nasopharyngitis (Infections and infestations) | 41 | 48
Urinary tract infection (Infections and infestations) | 26 | 8
Alanine aminotransferase increased (Investigations) | 64 | 6
Aspartate aminotransferase increased (Investigations) | 61 | 7
Blood alkaline phosphatase increased (Investigations) | 31 | 1
Blood lactate dehydrogenase increased (Investigations) | 22 | 1
Decreased appetite (Metabolism and nutrition disorders) | 47 | 25
Arthralgia (Musculoskeletal and connective tissue disorders) | 119 | 61
Back pain (Musculoskeletal and connective tissue disorders) | 38 | 34
Muscle spasms (Musculoskeletal and connective tissue disorders) | 39 | 13
Myalgia (Musculoskeletal and connective tissue disorders) | 70 | 40
Pain in extremity (Musculoskeletal and connective tissue disorders) | 60 | 38
Dizziness (Nervous system disorders) | 34 | 33
Dysgeusia (Nervous system disorders) | 29 | 12
Headache (Nervous system disorders) | 169 | 102
Cough (Respiratory, thoracic and mediastinal disorders) | 73 | 33
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 30 | 17
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 41 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 39 | 15
Alopecia (Skin and subcutaneous tissue disorders) | 24 | 18
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 54 | 10
Dry skin (Skin and subcutaneous tissue disorders) | 55 | 32
Erythema (Skin and subcutaneous tissue disorders) | 48 | 14
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 30 | 7
Night sweats (Skin and subcutaneous tissue disorders) | 23 | 11
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 24 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 40 | 29
Rash (Skin and subcutaneous tissue disorders) | 106 | 47
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 31 | 11
Hypertension (Vascular disorders) | 49 | 35
Lymphoedema (Vascular disorders) | 34 | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-05-31): https://cdn.clinicaltrials.gov/large-docs/83/NCT01682083/Prot_001.pdf
  • Statistical Analysis Plan (2017-05-31): https://cdn.clinicaltrials.gov/large-docs/83/NCT01682083/SAP_000.pdf